CLINICAL TRIAL: NCT02914418
Title: Feasibility Study to Investigate the Effects of Transcranial Magnetic Stimulation (TMS) Using Theta Burst Stimulation (TBS) to Treat Upper Limb Dysfunction and Spasticity in Patients With Spinal Cord Injury
Brief Title: Transcranial Magnetic Stimulation (TMS) for Upper Limb Dysfunction in Spinal Cord Injury: a Feasibility Study
Acronym: TUSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STH18997
Record Dates: First submitted 2016-08-23; First posted 2016-09-26 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Spinal Cord Injuries
Keywords: transcranial magnetic stimulation; Spinal Cord Injuries; Muscle Spasticity; Pain; Spinal Cord; Spinal Cord Diseases
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Spasticity; Pain; Spinal Cord Diseases | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active iTBS (Experimental): iTBS will be delivered using the 50Hz, 600 pulses protocol for 10 sessions over a period of two weeks. The hand representation of the primary motor cortex will targeted using a circular coil held over the vertex of skull. Intensity will be set to 80% of Resting Motor Threshold (RMT), which will be determined visually by the lowest percentage of stimulator output which can cause upper limb motor twitch in at least 5 out of 10 attempts.
  Interventions: Device: Transcranial Magnetic Stimulation using iTBS Paradigm
- Sham iTBS (Sham Comparator): Sham iTBS will be delivered using the 50Hz, 600 pulses protocol for 10 sessions over a period of two weeks. Intensity will be set at 80% RMT. Circular coil will be held over vertex of skull but angled away to ensure no neural stimulation.
  Interventions: Device: Transcranial Magnetic Stimulation using iTBS Paradigm

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation using iTBS Paradigm — TMS is a non-invasive, painless method of stimulating the central and peripheral nervous system. ITBS is a form of TMS which is delivered for ~200sec and can promote changes in neural activity.
  Other Names: repetitive Transcranial Magnetic Stimulation

SUMMARY:
This study will investigate how repetitive transcranial magnetic stimulation (TMS) using intermittent theta-burst stimulation (iTBS) paradigm affects sensorimotor dysfunction such as pain, spasticity, motor weakness and sensory loss. TMS is technique which allows non-invasive stimulation of the cortex, and can modulate activity of neurons. The purpose of this study will be to assess the feasibility of using TMS with iTBS paradigm to treat sensorimotor dysfunction in people with incomplete spinal cord injury affecting the upper limbs.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years old inclusive
* Traumatic and non-traumatic tetraplegic patient following chronic incomplete (AIS C or D) SCI injury (sustained at least three months ago)
* Referred to the Sheffield Spinal Injuries Centre
* Be able to provide written informed consent or verbal consent in the presence of an independent witness
* Spasticity affecting upper limbs with a Modified Ashworth scale (MAS) 2 or above
* Stable medical treatment for at least 1 week before and 1 week after TMS application
* Stable medical condition

Exclusion Criteria:

* Aged less than 18 years old
* Lack the mental capacity to consent
* Ventilated patients with sedation
* Very acute (<3 months) SCI patients
* Implanted electrical devices such as pacemakers, Concomitant neurological conditions, including any history of epilepsy
* Significant joint-related limitation of passive range of movement
* Unable to attend all TMS sessions
* Pregnancy
* Inability to tolerate TBS
* Significant upper limb contractures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Feasibility Criteria 1: Number of participants recruited | Through to study completion, up to 6 months
  Recruitment of 20 participants within 6 months (i.e. 3 - 4 participants per month)
Feasibility Criteria 2: Number of participants completing intervention protocol | Through to study completion, up to 6 months
  10 participants completing full intervention protocol
Feasibility Criteria 3: Number of Valid data sets | Through to study completion, up to 6 months
  10 complete valid data sets
Feasibility Criteria 4: Number of Serious Adverse Events Experienced by Participants | Through to study completion, up to 6 months
  No serious adverse events

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | Baseline and 2 weeks
  MAS is a clinical assessment of spasticity. Spasticity of wrist extensors, flexors, elbow extensors and flexors of both upper limbs will be assessed.
Range of Motion (RoM) | Baseline and 2 weeks
  Active RoM of wrist extension, flexion, elbow extension and flexion of both of both upper limbs will be measured using a goniometer.
Leeds Arm Spasticity Impact Scale (LASIS) | Baseline and 2 weeks
  Questionnaire assessing impact of spasticity on a person.
Visual Analogue Scale (Spasticity) (VAS-S) | Baseline and 2 weeks
  A 100mm line with two statements at each end (No spasticity, worst spasticity). The patient will mark on the line their own perception of how bad they feel their spasticity is.
American Spinal Injuries Association Impairment Scale (AIS) (Inc. grading, upper extremity motor score, lower extremity motor score, light touch and pin prick scores) | Baseline and 2 weeks
  A clinical assessment of sensory dermatomes and key muscle groups of upper and lower limbs.
Spinal Cord Independence Measure (SCIM) - Version 3 | Baseline and 2 weeks
  scale developed to address the ability of SCI patients to perform basic activities of daily living independently.
Visual Analogue Scale (Pain) - (VAS-P) | Baseline and 2 weeks
  A 100mm line with two statements at each end (no pain, worst pain). The patient will mark on the line their own perception of how bad they feel their pain is.

CONTACTS AND LOCATIONS:
Overall Officials: Ram Hariharan, MD, Study Chair — Sheffield Teaching Hospitals NHS Foundation Trust; Ali Gharooni, Principal Investigator — Sheffield Teaching Hospital NHS Foundation Trust. University of Sheffield.
Locations (1):
- Princess Royal Spinal Injuries Centre, Northern General Hospital., Sheffield, South Yourkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided